CLINICAL TRIAL: NCT01955317
Title: Waterless Hand Cleansing With Chlorhexidine During the Perinatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-13023
Record Dates: First submitted 2013-08-25; First posted 2013-10-07 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2016-08

CONDITIONS: Hand Washing Behavior; Hand Cleansing Behavior; Chlorhexidine; Neonatal Period
Keywords: Neonate; Bangladesh; Health behavior; Handwashing; Developing countries; Infectious disease
MeSH Terms: conditions — Health Behavior; Communicable Diseases | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chlorhexidine intervention (Experimental): The intervention arm will also receive hand hygiene counselling with chlorhexidine and a pump bottle with chlorhexidine lotion along with mothers and neonatal health counseling.
  Interventions: Behavioral: Hand cleansing with chlorhexidine
- Control (Active Comparator): This arm will receive maternal and neonatal health counselling which includes discussion and education about antenatal care, safe and clean delivery, recognition of danger signs for the mother and neonate, immediate new born care, and essential new born care. Each mother will receive a clean delivery kit and pictoral cue cards for danger sign recognition.
  Interventions: Behavioral: Mother and neonatal health counselling

INTERVENTIONS:
Behavioral: Hand cleansing with chlorhexidine — Pregnant women in the intervention arm will receive an intensive hand cleansing promotion delivered at 3 in-home visits between one month prenatal and 1 week post natal. The intervention will promote and discuss with mothers the benefits of hand cleansing with chlorhexidine before breastfeeding, before umbilical cord care, after contact with respiratory secretions, and the convenience of using a waterless hand sanitizer especially during the neonatal period. Each mother will receive a half-liter pump bottle with chlorhexidine lotion. The program will also educate mothers about infectious causes of morbidity and mortality in neonates and promote understanding of the risk to the neonate from these diseases.
  Arms: chlorhexidine intervention
Behavioral: Mother and neonatal health counselling — This arms will receive maternal and neonatal health counselling which includes discussion and education about antenatal care, safe and clean delivery, recognition of danger signs for the mother and neonate, immediate new born care, and essential new born care. Each mother will receive a clean delivery kit and pictoral cue cards for danger sign recognition.
  Arms: Control

SUMMARY:
Background (brief):

1. Burden:

   Neonatal death still unacceptably high in low income countries. The common causes of neonatal death are pneumonia, sepsis and omphalitis. Many neonatal infections occur because the mother's hands or the hands of the person who attended the birth are unclean. Our previous study found that there was substantial concern about excessive exposure of the mother or the neonate to water during handwashing because of the perception that frequent contact with water could lead to respiratory illness.
2. Knowledge gap:

   Chlorhexidine has been evaluated for use in hand hygiene applications in high-income countries, particularly in healthcare, but it has not been evaluated or promoted for hand cleansing at the household level in low- and middle-income countries.
3. Relevance:

A waterless hand cleanser employing chlorhexidine would overcome important barriers to handwashing with soap, perceptions of cold resulting from exposure to water, and the time limitations perceived by mothers.

Hypothesis: Mothers who are exposed to a chlorhexidine-based hand cleansing intervention will clean their hands (with chlorhexidine or soap and water) more frequently than mothers who are not exposed to the chlorhexidine-based hand cleansing program.

Objectives:

The primary objective

1. To demonstrate the behavioural impact of chlorhexidine-based hand hygiene intervention on hand cleansing of mothers during the neonatal period The secondary objectives
2. To demonstrate the impact of chlorhexidine-based hand hygiene intervention on hand cleansing of other family members, visitors to the neonate, and birth attendants during the neonatal period
3. To evaluate the acceptability of chlorhexidine for hand cleansing in the neonatal period among mothers, other family members, and birth attendants

Methods:

We propose a randomized controlled trial in a rural area of Bangladesh, with an active control. Randomization will be at the level of the participating pregnant woman. Each arm will include 150 participants. All intervention visits will follow baseline data collection. A trained health and hygiene promoter will carry out two visits in the antenatal period and one postnatal visit to deliver intervention messages.

Outcome measures:

1. Observed hand cleansing behavior of mother with chlorhexidine or soap and water at critical times.
2. Observed hand cleansing behavior of other household members and visitors to home with chlorhexidine or soap and water at critical times.

DETAILED DESCRIPTION:
Neonates (babies < 28 days old) die at unacceptably high rates (26deaths per 1000 live births) in many resource-limited countries, accounting for about 40% of deaths among all children under 5 years old. Infections such as pneumonia, sepsis, and omphalitis are common causes of neonatal death. Many neonatal infections occur because the mother's hands or the hands of the person who attended the birth are unclean. In Nepal, newborns who survived were significantly more likely than newborns who died to have mothers reporting handwashing, and birth attendants who were reported to wash hands before the delivery. But, mothers and birth attendants often do not wash their hands, despite the vulnerability of the neonatal period.

The traditional approach to improving handwashing among caregivers of young children is to teach about critical times to wash hands and how to wash hands. This narrow, prescriptive approach ignores the barriers to hand hygiene unique to the Perinatal and neonatal periods. Moreover, our qualitative findings suggest that frequent handwashing with water may not be acceptable. That is, both mothers and birth attendants reported that, when mothers come into contact with water frequently (e.g. by washing hands often), the newborn child is at risk of developing upper and lower respiratory infection. A novel technological solution - one that provides efficiency and portability and obviates the need for washing with water - may overcome important obstacles to improving hand cleansing behavior in the neonatal period.

During the discrete time frame of the neonatal period, chlorhexidine for hand cleansing represents a focused intervention with substantial potential for scalability. The shelf-life of chlorhexidine is long (2-3 years), facilitating its scaling up and efficient distribution, for example, in clean delivery kits that are provided to low-income mothers throughout resource-limited countries.

Given the potential for this low-technology solution to break through critical barriers to handwashing with water and soap, and markedly reduce neonatal mortality, we propose to conduct a randomized controlled trial to evaluate the impact of a chlorhexidine-based hand cleansing intervention on maternal, familial, and birth attendant hand cleansing behavior in the peripartum and neonatal periods.

Methods Study design

We propose a randomized controlled trial in a rural area of Bangladesh, with an active control. The two treatment arms are:

* Active control arm Maternal and neonatal health counseling (described in "Intervention" section)
* Intervention arm

  * Maternal and neonatal health counseling
  * Hand hygiene promotion (described in "Intervention" section) Randomization will be at the level of the participating pregnant woman (i.e. individual-level randomization). We will use a block randomization strategy to randomize participants to either the intervention or active control arm.

The intervention:

All intervention visits will follow baseline data collection. A trained health and hygiene promoter will carry out two visits in the antenatal period (at 34-35 weeks and at 36-38 weeks) and one postnatal visit (1-3 days after delivery) to deliver intervention messages.

Maternal and neonatal health counseling:

Study participants in both intervention and control arms will receive maternal and neonatal health counseling. The objectives of the maternal and neonatal health counseling are to:

* Highlight the vulnerability of the neonatal period
* Inform participant and her family of the schedule recommended by the Government of Bangladesh for prenatal care and strongly encourage participants to seek appropriate prenatal care, including Tetanus Toxoid vaccination. Tetanus toxoid is provided free of cost as part of antenatal care at all Government of Bangladesh health facilities.
* Discuss birth plans and encourage participants to develop a birth plan, including location of the birth, materials, persons needed and an emergency plan.
* Introduce and discuss the use of a clean delivery kit for hygienic delivery to reduce infections. This will include instructions on cutting the umbilical cord. Provide a clean delivery kit to the participant, which will include a clean blade, clean string for tying the cord, clean mat for the mother to lie on, among other items.
* Encourage close family members to motivate or demand hand washing with soap by birth attendants before and during labor and delivery.
* Discuss maternal danger signs with participant and her family and encourage care seeking when recognized
* Discuss neonatal danger signs with participant and her family and encourage care seeking when recognized
* Discuss neonatal hypothermia prevention with participant and her family and work with the family to build acceptance of the message
* Discuss the benefit of immediate and exclusive breastfeeding with participant and her family and work with the family to build acceptance of the message
* Provide chlorhexidine and gauze, and explain chlorhexidine cord care to the participant and work with her and her family.

Materials: Each participant will be given a clean delivery kit and a culturally appropriate pictorial card depicting each of the danger signs for the mother pre-, during, and post-labor, and for the neonate.

Description of behavioral communication approach: Interactions with the health and hygiene promoter will be in the form of a discussion where the health/hygiene promoter will facilitate discussions and provide explanation and guidance as needed.

Hand hygiene counseling:

Objectives of hand hygiene counseling:

* Present hand cleansing as an opportunity for the mother to protect the health of her child, and to improve perception of herself as a good mother
* Remind of the vulnerability of the newborn period, and suggest that the use of chlorhexidine for hand cleansing makes loving hands to be protective hands
* Encourage maternal self-efficacy for protecting the health of the baby
* Identify motivators and barriers to hand cleansing among mothers and other people that care for the baby
* Identify critical times for hand cleansing with chlorhexidine
* Increase individual and social (family/compound) expectations for hand cleansing among mothers and other caregivers
* Guide family to create solution for barriers to hand cleansing
* Introduce chlorhexidine as a product to help protect the baby's health, demonstrate use and discuss who, when and how to use it.
* Discuss demanding or motivating use of chlorhexidine by other family members, visitors and the birth attendant
* Set up a visual cue card, and a calendar with visual reminders in the home as references and cues for hand cleansing at specific critical times
* Discuss creating a habit of hand cleansing, what that concretely means and how to do so

Critical times for hand cleansing:

* For mothers and secondary caregivers:
* Before umbilical cord care
* After contact with respiratory secretions
* At three fixed times of day: morning, after lunch, and evening: given the residual antimicrobial effect of chlorhexidine, hand cleansing at these fixed times will result in hands being protected from contamination for much of the day.
* For visitors to the household and for children:
* Before touching the neonate
* After contact with respiratory secretions or contact with nasal or oral mucosa

Timing of intervention visits:

Respondents randomized to the intervention arm will receive one hand hygiene promotion during the second visit (at 36-38 weeks of gestation) prior to the review of the maternal and neonatal health counseling.

Chlorhexidine for hand cleansing: We are positioning chlorhexidine as a product that is of unique importance in the neonatal period, and may have substantive bactericidal and bacteriostatic effects, making it superior to soap for hand cleansing, particularly in the vulnerable newborn period.

Data collection Identification of pregnant women and selection criteria: The proposed study will be conducted in 4 unions in Mirzapur that are already under demographic surveillance. Pregnant women are routinely identified as part of the demographic surveillance.

Obtaining informed consent and baseline data collection: A data collector will describe the study to the pregnant woman at 32-34 weeks gestation and seek informed consent from her for participation. The data collector will also request informed consent from the head of household for interview of secondary caregivers regarding practices during the labor and delivery process, and two structured observations of hand cleansing behavior among all household members.

Randomization and initiation of intervention: We will use a block randomization strategy, using blocks of 4, to randomize participants to either the intervention or active control arm. Block randomization is also referred to as "restricted randomization" and allows for the numbers in the intervention arm to be roughly similar to those in the control arm throughout the enrolment period.

Objectives 1 and 2: Hand cleansing behavior measurement

To compare treatment arms with respect to mothers' hand cleansing behavior in the neonatal period (Objective 1), we will do the following:

1. Observe hand cleansing, either by use of chlorhexidine or by handwashing with water + soap, during 3-hour structured observations
2. Measure residual sanitizer weight and volume as markers of chlorhexidine consumption Structured observations involve the placement of a study staff member in the participant's home / household compound for an extended period of time in order to observe typical behaviors. In this study the observations will be conducted in both intervention and treatment arms by female field staff who will sit in a suitable place to observe the mothers without getting in the way of their normal care giving activities of the neonates. We are interested in observing the following behaviors during structured observations (Appendix 6).

Hand cleansing at critical times (either by chlorhexidine use or by washing hands with soap and water; handwashing with soap will be considered the corollary to chlorhexidine use since the control arm does not have access to chlorhexidine) Objective 3: Acceptability of chlorhexidine In both groups, we will record participant- or household member-initiated reporting of any skin reactions, other possible adverse events, and acceptability of the chlorhexidine with respect to ease of use, scent, skin comfort and the occurrence of skin reactions (Objective 3).

At approximately day 28 of the neonate's life, we will conduct an end line survey (Appendix 7) with the mother, during which we will assess the following in a quantitative manner in the intervention group:

* Acceptability of chlorhexidine
* Reported use of chlorhexidine versus handwashing hardware
* Behavioral determinants of hand hygiene We will collect qualitative data from a subset of mothers in the intervention arm to understand in-depth about barriers and motivators to chlorhexidine use for hand cleansing at the conclusion of all quantitative data collection.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women older than 18 years that are at 32-36 weeks gestation and intend to reside in the location which they are residing at the time of recruitment into the study through the remainder of the antenatal period and the first 4 weeks after birth.

Exclusion Criteria:

* Plans to move out of study area between enrollment and 1 month after birth.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Observed hand cleansing behavior of mother with chlorhexidine or soap and water at critical times | 1 week and one month after birth
  We will observe hand cleansing behavior of mother through 3 hours structured observations.

SECONDARY OUTCOMES:
Observed hand cleansing behavior of other household members and visitors to home with chlorhexidine or soap and water at critical times | 1 week and one month after birth
  We will observe hand cleansing behavior at critical time of other household members through 3 hours structured observations.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirzapur, Tāngāil, Dhaka Division, Bangladesh